CLINICAL TRIAL: NCT01560728
Title: Bringing What Works to Youth in Prison: An Evidence-Based Trauma Intervention
Brief Title: Bringing What Works to Youth in Corrections: A Trauma Intervention
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34MH095210-01 (NIH); 1R34MH095210-01 (NIH)
Record Dates: First submitted 2012-03-19; First posted 2012-03-22 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Post Traumatic Stress Disorder; Major Depressive Disorder; Dysthymia; Generalized Anxiety Disorder; Social Phobia; Panic Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Dysthymic Disorder; Generalized Anxiety Disorder; Phobia, Social; Panic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trauma-Focused CBT (Experimental): Adapted or modified Trauma-Focused Cognitive Behavioral Therapy
  Interventions: Behavioral: Trauma-Focused Cognitive Behavioral Therapy
- Wait list (No Intervention): Monitored while waiting for intervention

INTERVENTIONS:
Behavioral: Trauma-Focused Cognitive Behavioral Therapy — Individual psychotherapeutic approach occurring once per week for 12 to 20 weeks
  Arms: Trauma-Focused CBT

SUMMARY:
Youth with mental illnesses are disproportionately represented in juvenile correctional facilities and limited evidence exists about effective treatments in this setting. This study will adapt Trauma-Focused Cognitive Behavioral Therapy (TF-CBT), a treatment found to be efficacious in community settings, to the correctional setting and study the feasibility of its implementation. Conducted within Texas youth correctional facilities, the findings will be rapidly disseminated in the state. The goal is to enhance the TF-CBT approach to meet the unique needs of incarcerated youth and the correctional system, one of the priorities outlined in the National Institute of Mental Health Strategic Plan.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of one or more significant traumatic life events
* Current diagnosis of one of the following:

  * Post Traumatic Stress Disorder
  * Major Depressive Disorder
  * Dysthymia
  * Generalized Anxiety Disorder
  * Social Phobia
  * Panic Disorder
* Trauma symptom severity scores of 25 or greater.

Exclusion Criteria:

* Expected release date or transfer date within 5 months from study enrollment date
* Current inclusion in the Sex Offender Treatment Program
* Intellectual Quotient (IQ) less than 70
* Current high risk of suicidality
* Current symptoms of active psychosis

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2012-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Rate of change in UCLA PTSD Reaction Index (UCLA PTSD RI) Trauma Symptom Severity | Participants will be assessed at baseline and every 2 weeks for an average of 6 months
  Reduction in traumatic stress symptom severity

SECONDARY OUTCOMES:
Rate of change in Child Behavioral Checklist Youth Self-Report Total Score | Participants will be assessed at baseline and every 2 weeks for an average of 6 months
  Reduction in self-reported emotional and behavioral problem scores

CONTACTS AND LOCATIONS:
Overall Officials: Molly M Lopez, Ph.D., Principal Investigator — University of Texas at Austin
Locations (3):
- United States (3):
  - Ron Jackson State Juvenile Correctional Facility, Brownwood, Texas
  - Giddings State School, Giddings, Texas
  - McClennan County State Juvenile Correctional Facility, Mart, Texas